CLINICAL TRIAL: NCT06729853
Title: A Phase 1, Open-Label, Parallel-Group, Single-Dose Adaptive Study to Evaluate the Safety and Pharmacokinetics of SAP-001 in Adult Subjects With Normal and Impaired Renal Function
Brief Title: PK and Safety Evaluation Study of SAP-001 in Adult Subjects With Normal and Impaired Renal Function
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanton Pharma Pte. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SAP-001-104
Record Dates: First submitted 2024-12-04; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Gout; Hyperuricemia
MeSH Terms: conditions — Gout; Hyperuricemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Mild renal impairment (Experimental): Subjects with mild renal impairment
  Interventions: Drug: SAP-001
- Moderate renal impairment (Experimental): Subjects with moderate renal impairment
  Interventions: Drug: SAP-001
- Severe renal impairment (Experimental): Subjects with severe renal impairment(Optional)
  Interventions: Drug: SAP-001
- Healthy match (Experimental): Matched healthy subjects with normal renal function
  Interventions: Drug: SAP-001

INTERVENTIONS:
Drug: SAP-001 — a single oral dose of SAP-001

SUMMARY:
This is a multicenter, open-label, non-randomized, parallel-group, single-dose, 2-part, adaptive study in which up to approximately 32 adult subjects will be enrolled in one of 4 groups (8 subjects per group) with varying degrees of renal function.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

1. Provision of signed and dated informed consent form (ICF)
2. Subject is, as stated and in the opinion of the Investigator, willing and able to comply with the study drug regimen and all other protocol and study procedures and requirements, and is available for the duration of the study
3. Adult male or female
4. Subject is willing to comply with the contraceptive requirements as defined in APPENDIX 6
5. Aged at least 18 years but not older than 80 years
6. BMI ≥ 18.5 kg/m2 and < 42.0 kg/m2 at the time of Screening.
7. Light-, non- or ex-smoker (A light smoker is defined as someone using 10.0 nicotine units [1 unit = 1 cigarette] or less per day for at least 90 days prior to study drug administration. An ex-smoker is defined as someone who completely stopped using nicotine products for at least 180 days prior to study drug administration)
8. Having suitable venous access for blood sampling

   Subjects with Normal Renal Function (Group 4):
9. Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on the laboratory tests, physical examination (including vital signs) and/or ECG, as determined by an Investigator
10. Normal renal function with estimated glomerular filtration rate (eGFR) ≥ 90 mL/minute at Screening
11. Must match to the pooled mean age (± 10 years), BMI (within 20%) and sex (ratio should be similar) of mild, moderate (if applicable), and severe (if applicable) renal impaired subjects

    Subjects with mild, moderate, or severe renal impairment (Groups 1, 2 and 3, respectively):
12. Considered clinically stable in the opinion of an Investigator
13. Presence of mild renal impairment (eGFR ≥ 60 and < 90 mL/min), moderate renal impairment (eGFR ≥ 30 and < 60 mL/min) or severe renal impairment (eGFR≥ 15 and < 30 mL/min) at Screening. Renal impairment should be stable for at least 1 month prior to Screening (change in eGFR should not be more than 25%).

Note: The Investigator can order a repeat of eGFR if it is determined that the initial value is inconsistent with the historical values for a particular subject

Exclusion Criteria:

All subjects:

1. Female who is lactating
2. Female who is pregnant according to the pregnancy test at Screening or prior to study drug administration
3. History of significant hypersensitivity to SAP-001 or any related products (including excipients of the formulation) as well as severe hypersensitivity reactions (like angioedema) to any drugs
4. Positive screening results to HIV Ag/Ab Combo and Hepatitis B surface antigen (HBsAg)
5. Positive reflex test for Hepatitis C antibody (positive Hepatitis C antibody is allowed if HCV RNA is not detected)
6. Presence or history of any disorder that could interfere with completion of the study based on the opinion of an Investigator
7. Intake of SAP-001 or any Investigational Product (IP) in the 28 days (or 5 times the half-life of the drug, whichever is longer) prior to study drug administration
8. Have urinary incontinence without catheterization
9. Reception of blood products within 3 months prior to study drug administration
10. Donation of 50 mL or more of blood in the 28 days prior to Screening
11. Donation of 500 mL or more of blood within 56 days prior to Screening.
12. Donation of plasma within 2 weeks prior to Screening or platelets within 6 weeks prior to Screening
13. Inclusion in a previous group for this clinical study

    Subjects with Normal Renal Function (Group 4):
14. Presence of significant gastrointestinal, liver, or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs or known to potentiate or predispose to undesired effects
15. History of significant gastrointestinal, liver or kidney disease that may affect drug bioavailability
16. Presence of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
17. Presence of out-of-range cardiac interval (eg, QTcF > 440 msec) based on the mean of the triplicate ECG values at Screening or other clinically significant ECG abnormalities, unless deemed non-significant by an Investigator
18. Positive test result for alcohol and/or drugs of abuse at Screening or prior to study drug administration
19. Seated blood pressure below 90/60 mmHg at Screening and prior to dosing
20. Seated blood pressure higher than 140/90 mmHg at Screening and prior to dosing
21. Seated pulse rate less than 40 beats per minutes (bpm) or more than 100 bpm at Screening and prior to dosing
22. Any clinically significant illness in the 28 days prior to study drug administration
23. Use of any prescription drugs (with the exception of hormonal contraceptives or hormone replacement therapy) in the 28 days prior to study drug administration that, in the opinion of an Investigator, would put into question the status of the participant as healthy
24. Use of St. John's wort in the 28 days prior to study drug administration
25. Use of over-the-counter drugs and natural health products (eg, herbal remedies) in the 14 days (or 5 times the half-life of the drug, whichever is longer) prior to study drug administration
26. Use of any enzyme-modifying drugs, or drugs with effects on membrane transporters, including any strong cytochrome P450 3A4 and P-glycoprotein inducers and inhibitors in the previous 28 days prior to study drug administration

    Subjects with Renal Impairment (Groups 1, 2 and 3):
27. History of renal transplant
28. Seated blood pressure below 100/50 mmHg at Screening and prior to dosing
29. Seated blood pressure higher than 180/100 mmHg at Screening and prior to dosing
30. Seated pulse rate less than 50 bpm or more than 110 bpm at Screening and prior to dosing
31. History or presence, in the opinion of an Investigator, of significant clinically unstable respiratory, cardiovascular, pulmonary, hepatic, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease
32. Presence of poorly controlled Type 1 or Type 2 diabetes as defined by hemoglobin A1c > 10%
33. Presence of clinically significant physical examination, laboratory test, or ECG finding that, in the opinion of an Investigator and/or Sponsor, may interfere with any aspect of study conduct or interpretation of results
34. Subjects requiring treatment for renal impairment or other chronic disease (eg, well-controlled diabetes, hypertension) must be on a stable treatment plan (medicines, doses, and regimens) for at least 14 days (except insulin) prior to study drug administration and during the entire study. Small adjustments in the dosages of some concomitant medications may be permitted during the study and will be discussed on a case-by-case basis. In all cases, the subjects' treatment history must be reviewed and their enrollment must be agreed to by both an Investigator and the Sponsor's Medical Monitor
35. Positive screening of alcohol and/or drugs of abuse at Screening or prior to study drug administration unless results can be explained by a prescription medication
36. Concurrent use of medications known to affect the elimination of serum creatinine (eg, trimethoprim/sulfamethoxazole [Bactrim®] or cimetidine [Tagamet®]) and competitors of renal tubular secretion (eg, probenecid) within 30 days prior to study drug administration or anticipated need for these therapies through to the last PK sample of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2025-01-17 (Estimated); Study Completion 2025-04-28 (Estimated)

PRIMARY OUTCOMES:
maximum observed concentration (Cmax) | day 8
  The primary PK endpoints
AUC from time 0 to time of last quantifiable sample (AUC0-T) | day 8
  The primary PK endpoints
apparent clearance (CL/F) | day 8
  The primary PK endpoints

SECONDARY OUTCOMES:
time to maximum concentration (Tmax) | day 8
  Plasma PK parameters
AUC from time 0 extrapolated to infinity (AUC0-∞) | day 8
  Plasma PK parameters
terminal elimination half-life (Thalf) | day 8
  Plasma PK parameters
volume of distribution (Vz/F) | day 8
  Plasma PK parameters
Ae(0-T) (amount excreted) | day 8
  Urine PK parameters:
Fraction of dose excreted in urine (fe) | day 8
  Urine PK parameters:
CLr (renal clearance) | day 8
  Urine PK parameters:

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Genesis Clinical Research, Tampa, Florida
  - Nucleus Network Pty Ltd, Saint Paul, Minnesota